CLINICAL TRIAL: NCT04790448
Title: A Phase Ia/II, Single Arm Trial on the Efficacy of Vemurafenib in Combination With Irinotecan and Cetuximab in BRAF V600E-Mutant Metastatic Colorectal Cancer
Brief Title: Efficacy of VIC Regimen in BRAF Mutant Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIC-BRAFMT-mCRC
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Cetuximab; Irinotecan; Vemurafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIC regimen (Experimental): Patients will receive VIC regimen every 2 weeks:
  Cetuximab 500mg/m2 IV on Day 1; Irinotecan 180mg/m2 IV on Day 1 (If patient carries UGT*28 7/7 or UGT*6 A/A or UGT*28 6/7 and UGT*6 A/G variants, use Irinotecan IV 150mg/m2 instead); Vemurafenib PO BID on Days 1 to 14 (Dosage: 480mg; 720mg; 960mg, determined by the maximum tolerated dose (MTD) in Phase Ia trial).
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cetuximab — Route of administration: Intravenous
  Other Names: C225; Erbitux
Drug: Irinotecan — Route of administration: Intravenous
  Other Names: CPT-11; Camptothecin-11; Camptosar
Drug: Vemurafenib — Route of administration: Oral
  Other Names: Zelboraf

SUMMARY:
This prospective, multicenter, single arm clinical trial was designed to evaluate the efficacy and safety of Vemurafenib in combination with Irinotecan and Cetuximab in the treatment of BRAF V600E-Mutant Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To evaluate the Overall Response Rate (ORR) of v-raf murine sarcoma viral oncogene homolog B (BRAF) V600E mutant metastatic colorectal cancer patients treated with Vemurafenib in combination with Irinotecan and Cetuximab (VIC regimen).

SECONDARY OBJECTIVES:

To evaluate the Progression Free Survival (PFS), Overall Survival (OS), safety and toxicity of VIC regimen in the treatment of BRAF V600E mutant colon cancer.

EXPLORATORY OBJECTIVES:

Mechanism of primary and secondary resistance to VIC regimen in the treatment of BRAF V600E mutant colon cancer.

OUTLINE:

Patients receive Cetuximab and Irinotecan intravenously on day 1 and Vemurafenib orally (PO) twice daily (BID) on days 1 to 14. Courses are repeated every 2 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic colorectal cancer
* Histopathological or ctDNA analysis positive for BRAF V600E mutant
* Patients must have had at least undergone one first line treatment with FOLFOX or FOLFIRI or FOLFOXIRI±Bevacizumab before disease progression.
* Measurable and assessable disease according to RECIST 1.1 criteria
* Adequate hematologic function (Platelet>90×109/L; White blood cells>3.0×109/L; Neutrophils>1.5×109/L; Hb>10.0g/100ml)
* Serum bilirubin ≤1.5 times the upper limit of normal (ULN), transaminase ≤5 times ULN
* No ascites, normal coagulation function, albumin ≥35g/L
* Child-Pugh class A
* Serum creatinine is less than the upper limit of normal (ULN), or calculated creatinine clearance rate> 50ml/min (using Cockcroft-Gault equation)
* ECOG performance status of grade 0-2
* Life expectancy> 3 months
* Patients must provide a signed Informed Consent Form
* Patients must have good compliance till the end of this study

Exclusion Criteria:

* Patients with KRAS and NRAS mutations
* Previously received anti-EGFR monoclonal antibodies or EGFR inhibitors, BRAF inhibitors (with the exception of regorafenib)
* Patients with known contraindications to receiving cetuximab or irinotecan at the planned dose
* Patients with retinal vein occlusion or have current risk factors for retinal vein occlusion (for example, uncontrolled glaucoma or ocular hypertension)
* History of acute or chronic pancreatitis
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive drugs or surgery) within 12 months prior to enrollment
* Gastrointestinal diseases that may greatly affect the absorption of Vimurafenib (for example, ulcer disease, uncontrolled vomiting, malabsorption syndrome, small bowel resection and reduced intestinal absorption)
* Neuromuscular diseases associated with elevated CK (eg, inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Patients with any residual CTCAE ≥ Grade 2 toxicity from previous anti-tumor therapy (excluding hair loss or neuropathy of Grade 2 and above)
* History of HIV infection
* Active hepatitis B or C infection
* History of Gilbert syndrome
* Interstitial pneumonia or widespread symptomatic interstitial pulmonary fibrosis
* Serious uncontrollable systemic complications such as infection or diabetes
* Clinically serious cardiovascular diseases such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), hypertension that cannot be controlled after proper medical treatment, unstable angina pectoris, congestion Heart failure (NYHA 2-4), arrhythmia requiring medication
* History of or showing signs of a central nervous system disease (such as primary brain tumors, epilepsy that cannot be controlled by standard treatment, any brain metastases or history of stroke)
* Patients must not suffer from other uncontrolled concurrent diseases, including but not limited to hypertensive crisis or hypertensive encephalopathy, active bleeding, uncontrolled infections/diseases, uncontrolled non-malignant medical diseases or use research therapies that could worsen non-malignant medical diseases or mental illnesses/social conditions
* No history of other malignant tumors in the past 5 years (excluding skin basal cell carcinoma and/or cervical carcinoma in situ and/or thyroid cancer after radical resection)
* Patients allergic to any drugs in the study
* Patients must not be pregnant or breastfeeding
* Women of reproductive potential (<2 years after the last menstruation) who have not used or refused to use effective non- hormonal contraceptive methods (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or sterilization) or Men wanting to keep their reproductive potential.
* Patients unable or unwilling to comply with the protocol of this clinical trial
* Existence of any other diseases, dysfunction caused by metastatic lesions, or suspicious diseases found during physical examination, which may indicate contraindications to the use of the drugs in this study or could bring about high risk of treatment-related complications to the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate from the date of first drug administration until the date of first documented progression or date of death, whichever came first. | up to 17 months
  The proportion of patients who achieved a complete or partial response as their best overall response based on RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression free survival from the date of first drug administration until the date of first documented progression or date of death, whichever came first. | up to 17 months
  The length of time during and after the treatment of the disease, that a patient lives with the disease without its aggravation
Overall Survival from the date of first drug administration until the date of death from any cause. | up to 17 months
  The length of time from the start of treatment that patients diagnosed are still alive
Number of patients with adverse events and severity according to NCI CTCAE v5.0 | up to 6 months
  Summary of the Adverse events experienced during treatment related to the drug used in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided